CLINICAL TRIAL: NCT01747889
Title: Objective and Subjective Outcomes of an Electronic Chest Drainage System Versus Traditional Devices: a Randomized Comparison
Brief Title: Objective and Subjective Outcomes of an Electronic Chest Drainage System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedali Riuniti Ancona (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other); The University of Hong Kong (Other); Yale University (Other)
Responsible Party: Principal Investigator, Cecilia Pompili, MD, Ospedali Riuniti Ancona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PATSAT-2012-1
Record Dates: First submitted 2012-12-07; First posted 2012-12-12 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Lung Cancer
Keywords: chest tube; lung resection; patient satisfaction; mobility
MeSH Terms: conditions — Lung Neoplasms; Patient Satisfaction

ARMS (2):
- Electronic system (Experimental): patients managed with an electronic chest drainage system
  Interventions: Device: electronic chest drainage system
- traditional system (No Intervention): patients managed with a traditional analogue chest drainage system

INTERVENTIONS:
Device: electronic chest drainage system — Patients in the intervention arm are connected to Thopaz, electronic drainage system immediately after closure of the chest, patients in the control group are connected to a traditional system. Chest tubes in both groups are then connected to suction of -20 cmH2O and maintained at that level until post-operative day #1.
  On the morning of post-operative day #1, presence of air leak will be recorded on suction. Then, suction will be decreased to -8 cmH2O (so-called water seal). At that time, management of chest tube drainage and decision for chest tube removal will be dictated by clinical signs, symptoms, and surgeon preference following the standard clinical algorithm for post-operative care of general thoracic patients
  Arms: Electronic system

SUMMARY:
This study is designed to compare the Thopaz chest tube drainage system to the traditional collection chamber system. The Thopaz system is already in clinical use in the United States and throughout the world. As such, this study is not evaluating safety or efficacy of this system both of which have already been demonstrated. This study's primary aim is to determine whether the use of a digital chest drainage system compared with a traditional system affects duration of chest drainage and length of hospital stay.

Furthermore, we aim to determine whether the use of a digital chest drainage system compared with a traditional system increases the total distance of ambulation in the first 48 hours after thoracic surgery and affects overall patient satisfaction in the peri-operative period.

Finally, we want to determine whether the aforementioned outcomes relative to the chest tube drainage systems differ in different parts of the world.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to read, understand, and provide written Informed Consent
2. Age range of 18-90 years
3. Patients undergoing a segmentectomy, lobectomy, or bilobectomy. Both open and minimally invasive (thoracoscopic or robotic) resections are acceptable.

Exclusion Criteria:

1. Patients unstable enough to require ICU care upon completion of the resection
2. Redo thoracotomies

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Duration of chest tubes | date of chest tube removal

SECONDARY OUTCOMES:
total distance of ambulation in the first 48 postoperative hours | 48 hours after surgery

OTHER OUTCOMES:
overall patient satisfaction with chest drainage system. | 48 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Pompili, MD, Principal Investigator — Ospedali Riuniti Ancona, Italy
Locations (1):
- Ospedali Riuniti Ancona, Ancona, Italy

REFERENCES:
- [Derived] Pompili C, Detterbeck F, Papagiannopoulos K, Sihoe A, Vachlas K, Maxfield MW, Lim HC, Brunelli A. Multicenter international randomized comparison of objective and subjective outcomes between electronic and traditional chest drainage systems. Ann Thorac Surg. 2014 Aug;98(2):490-6; discussion 496-7. doi: 10.1016/j.athoracsur.2014.03.043. Epub 2014 Jun 4. PMID 24906602